CLINICAL TRIAL: NCT04575779
Title: Evaluation of the Clinical Outcome of Cyclosporine Short Infusion Versus Continuous Infusion Post Allogenic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Shaymaa Mohammed El-Awady (Other)
Responsible Party: Sponsor-Investigator, Shaymaa Mohammed El-Awady, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: 70
Record Dates: First submitted 2020-09-19; First posted 2020-10-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Allogenic Bone Marrow Transplantation
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Cyclosporin of a daily dose of 3 mg/kg/day intravenously over 2 h (short infusion) every 12 h
  Interventions: Drug: Cyclosporin with a daily dose of 3 mg/kg/day intravenously over 2 h (short infusion) every 12 h
- Group B: Administer cyclosporin daily dose of 3 mg/kg/day in a continuous infusion over 23 h every 24 h.
  Interventions: Drug: Cyclosporin with a daily dose of 3 mg/kg/day intravenously over 2 h (short infusion) every 12 h

INTERVENTIONS:
Drug: Cyclosporin with a daily dose of 3 mg/kg/day intravenously over 2 h (short infusion) every 12 h — To determine whether administering CsA at a dailydose of 3 mg/kg/day intravenously(i.v.) in 2 hrs (short infusion) twice-daily will achieve C2 blood levels of at least 800 mg/l and whether it will be feasible and safe or not.

SUMMARY:
This study focuses on the basis for current immunosuppressive strategies in patients undergoing allogeneic haematopoietic stem cell transplantation at the bone marrow transplantation unit in Ain Shams university hospitals. It discusses whether there is room for improving both the monitoring and the delivery of pharmacologically mediated immunosuppression in this population of patients. Our study will try to determine whether CsA administration at a daily dose of 3 mg/kg/day intravenously (IV) in 2 hrs (short infusion) twice-daily will achieve C2 blood levels of at least 800 mg/l and whether it will be feasible and safe or not.

DETAILED DESCRIPTION:
Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) is considered as a curative treatment for patients with haematological malignancies like leukaemia, myelodysplasia, lymphoma, and multiple myeloma. However, graft-versus-host disease (GvHD) both in its acute and chronic forms, has limited the benefits of allogeneic HSCT by significant morbidity and mortality.

Pharmacological suppression of the donor-derived alloreactive immune response has played a central role in reducing the morbidity and mortality of graft-versus-host disease (GvHD), which remains the major cause of toxicity after allogeneic stem cell transplantation (SCT).

Graft versus host disease (GvHD) is a condition that might occur after an allogenic transplant, In GvHD, the donated bone marrow or peripheral blood stem cells view the recipient's body as foreign, and the donated cells/bone marrow attack the body. There are two forms of GvHD: Acute graft versus host disease (aGvHD) and Chronic graft versus host disease (cGvHD). As an allogeneic transplant recipient, the patient might experience either form of GvHD, both forms, or neither.

Acute GvHD, which results from an interaction of donor T lymphocytes with the recipient's antigens, occurs in approximately 30%-60% of patients after allogeneic Hematopoietic Stem Cell Transplantation (HSCT). At the same time, it has become clear that the intensity of post-transplant immunosuppression is one of the most important determinants of relapse risk through its impact on the potency of an immunologically mediated graft-versus leukaemia (GVL) effect.

Among the variety of immunosuppressants available, cyclosporin A (CsA) has been the most extensively used drug to prevent or treat graft-versus-host disease (GvHD) in hematopoietic stem cell transplant (HSCT) recipients, since its introduction in the 1970s. It has been shown that CsA is effective in preventing and controlling acute and chronic GvHD.

Cyclosporine is an immunosuppressive agent, a metabolite extracted from the fungus Tolypocladium. It is a potent suppressor of the immune system, particularly T-lymphocytes. Cyclosporine binds to the intracellular receptor cyclophilin, subsequently inhibiting cytokine production, including interleukin-2 and 4, tumour necrosis factor-alpha, and interferon-gamma, which leads to impairment of normal lymphoid cell activation.

Other mechanisms may contribute to immunosuppression. Cyclosporine is cell cycle phase-specific; lymphocytes in the G0 or G1 phase of the cell cycle are specifically and reversibly inhibited. Direct cytotoxic effects on T- and B-lymphocytes have also been demonstrated.

The cyclosporine (CsA) acts in a concentration-dependent rather than a time-dependent fashion. It has been shown that the most significant pharmacodynamic effect occurs within the first two h of exposure (C2) at peak CsA levels of 800-2285 mg/l which result in 70-96% calcineurin inhibition and maximum suppression of IL-2 release from T cells.

Pharmacokinetics of cyclosporine (CsA) is highly complex and affected by many factors like demographics, concurrent medications and type of primary disease for which transplantation was indicated. Moreover, the complexity of CsA pharmacokinetics is increasing in critically ill patients in acute post-transplantation phase due to the presence of additional several clinical factors simultaneously affecting the in-vivo behaviour of CsA. This made very little research investigating the pharmacokinetic behaviour of CsA in acute post-transplantation period.

This study will focus on the basis for current immunosuppressive strategies in patients undergoing allogeneic haematopoietic stem cell transplantation at the bone marrow transplantation unit in Ain Shams university hospitals and discuss whether there is room for improving both the monitoring and the delivery of pharmacologically mediated immunosuppression in this population of patients.

Although it has already been known that the clinical effect of the cyclosporine (CsA) depends on the reached concentration levels in the blood, the best way of therapeutic monitoring of this drug is not universally accepted. The measurement of the drug concentration. level in the blood prior to the administration of the next successive dose (C0) and dosing of the drug on the basis of this drug concentration, represents the more common way of CsA therapeutic monitoring. Recently, it has been shown that C0 does not correlate well with the episodes of acute rejection, and undesirable drug effects as well.

Many studies showed that the absorption, but not the elimination phase, is primarily significant for the cyclosporine (CsA) effectiveness and that the area under the concentration-time curve in the first 4 hours after the drug administration (AUC0-4) adequately reflects the exposure of the organism to the drug and correlates well with clinical events. It was also shown that out of all drug concentration levels separately measured at some points of time during the absorption phase; the drug concentration level determined 2 hours after the administration (C2) correlates the best with the area under the concentration-time curve in the first 4 hours after the drug administration (AUC0-4).

In the past few years, considerable refinement has occurred in the pharmacologically mediated immunosuppressive strategies utilized in recipients of solid organ transplants. This has occurred through the use of more precise methods of monitoring established agents, principally cyclosporin (CsA), which have been shown to reduce the risk of graft rejection in the setting of both kidney and liver transplantation. This experience suggests that there may be scope for translating the advances that have been made in the field of solid organ transplantation to recipients of allogeneic haematopoietic stem cells.

The drug concentration level determined 2 hours after the administration (C2) monitoring has been adopted for renal, liver and heart transplant recipients as the two h peak concentration correlates well with the area under the concentration-time curve (AUC) from 0 to 4 h after giving the drug and that this predicts the occurrence of acute rejection and nephrotoxicity.

The drug concentration level determined 2 hours after the administration (C2) monitoring is also associated with clinical benefits as a reduction in graft rejections after solid organ transplantation. Amazingly, data on pharmacokinetics and target C2 levels are lacking in Hematopoietic Stem Cell Transplantation (HSCT) patients. Moreover, there is no consensus about how cyclosporin (CsA) should be administered with some centres giving 1 or 2 intermittent infusions and others continuous 24 h infusion. Hence, our study will try to determine whether administering CsA at a daily dose of 3 mg/kg/day intravenously(i.v.) in 2 hrs (short infusion) twice-daily will achieve C2 blood levels of at least 800 mg/l and whether it will be feasible and safe or not.

ELIGIBILITY:
Inclusion Criteria:

* Adult ages >18 years.
* Patients undergoing allogeneic stem cell transplantation, matched or mismatched related donors.
* Had never been exposed to cyclosporin before.

Exclusion Criteria:

* Patients with a hypersensitivity to cyclosporin or to any of the ingredients of the formulation.
* Patient with abnormal hepatic functions.
* Patient with abnormal renal functions with elevated serum creatinine levels in excess of 220 mmol/l at study entry.
* Patient receiving systemically active azoles within 2 weeks before Hematopoietic Stem Cell Transplantation (HSCT) patients.
* Patient with body mass index (BMI) above 30 kg/m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with related allogeneic stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Recording the occurrence of graft-versus-host disease (GvHD) events [Safety and tolerability] | Three months following transplantation date
  To compare between the administration of twice-daily cyclosporin infusion over two hours versus continuous cyclosporin infusion via recording the occurrence of graft-versus-host disease (GvHD) events
Recording the occurrence of cyclosporine toxicity adverse events [Safety and tolerability] | Three months following transplantation date
  To compare between the administration of twice-daily cyclosporin infusion over two hours versus continuous cyclosporin infusion via recording the occurrence of cyclosporine toxicity adverse events

SECONDARY OUTCOMES:
Recording the achievement of C2 (The drug concentration level determined 2 hours after the administration) blood levels of at least 800 mg/l. [Efficacy] | From Transplantation date till 3 months afterward
  Recording the patient success to achieve C2 (The drug concentration level determined 2 hours after the administration) blood levels of at least 800 mg/l.
Correlation with the the area under the concentration-time curve in the first 4 hours after the drug administration (AUC0-4) | From Transplantation date till day 8 afterward
  To determine which of the individual concentrations in the early phase after cyclosporin short infusion over 2 hours shows the best correlation with the the area under the concentration-time curve in the first 4 hours after the drug administration (AUC0-4).

CONTACTS AND LOCATIONS:
Locations (1):
- Shaymaa Mohammed Mohammed Youssef El-Awady, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Derived] El-Awady SMM, El Afifi AM, Afifi R, Sabri NA, Ahmed MA. Evaluation of the Clinical Outcomes of Cyclosporine Short Infusion Versus Continuous Infusion Postallogenic Stem Cell Transplantation. Eur J Drug Metab Pharmacokinet. 2025 Jan;50(1):53-64. doi: 10.1007/s13318-024-00927-y. Epub 2024 Nov 27. PMID 39601981